CLINICAL TRIAL: NCT01634035
Title: Correlation Between Glycated Hemoglobin and Mean Plasma Glucose in Hemodialysis Patients.
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 09-001; 09-001 (Other Grant/Funding Number: SIUH IRB)
Record Dates: First submitted 2010-06-03; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: ESRD
Keywords: glycated hemoglobin; mean plasma glucose
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Biospecimen Retention: None Retained — review of previous blood tests
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diabetic hemodialysis: all patient diabetic and on hemodialysis were involved if they are on hemodialysis for more than 3 months

SUMMARY:
The investigators are studying the correlation between Hba1c and the mean plasma glucose in diabetic hemodialysis patients.We are reviewing if HbA1c is a good clinical tool to assess glycemic control over a 3 months duration in hemodialysis patients

DETAILED DESCRIPTION:
The Hb turnover in hemodialysis population is higher than the general population leading to a general believe that HbA1c tend to underestimate mean plasma glucose.

The investigators are trying to define the correlation between mean plasma glucose and HbA1c in the hemodialysis population and trying to study the factors that could affect this correlation (dose of erythropoetin, ret count..) We are trying to see if HbA1c is a better tool to assess glycemic control over 1 month than glycemic control over 3 month.

This clinicaly will translate in obtaining HbA1c more frequently in hemodialysis patients to assess their glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Hemodialysis and diabetic
* Lab data are available for more than 6 months

Exclusion Criteria:

* Lab data not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all hemodialysis and diabetic population
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Measure levels of plasma blood glucose and HbA1c | 6 month intervals

SECONDARY OUTCOMES:
Measure ferritin, erythropoetin dose, reticulocytes count | 6 month intervals

CONTACTS AND LOCATIONS:
Overall Officials: suzanne el-sayegh, md, Principal Investigator — statenisland university hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States